CLINICAL TRIAL: NCT02987855
Title: Use of Autologous Adult Adipose-Derived Stem/Stromal Cells in Reflex Sympathetic Dystrophy (RSD), Complex Regional Pain Syndrome (CRPS), and Fibromyalgia
Brief Title: Adipose Stem/Stromal Cells in RSD, CRPS, Fibromyalgia
Acronym: ADcSVF-CRPS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn [COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform]
Sponsor: Healeon Medical Inc (Industry)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Science, Healeon Medical Inc
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSD-CRPS
Record Dates: First submitted 2016-12-05; First posted 2016-12-09 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: RSD (Reflex Sympathetic Dystrophy); CRPS - Complex Regional Pain Syndrome Type I; Fibromyalgia
MeSH Terms: conditions — Complex Regional Pain Syndromes; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipoaspiration Arm 1 (Experimental): Acquisition of Adipose-Derived tissue Stromal Vascular Fraction (AD-tSVF) via closed syringe lipoaspiration harvest of subdermal fat
  Interventions: Procedure: Lipoaspiration
- AD-cSVF Arm 2 (Experimental): ADcSVF Isolation of cellular stem/stromal cells from subdermal adipose-derived cellular stromal vascular fraction
  Interventions: Procedure: ADcSVF isolation
- Normal Saline IV Arm 3 (Experimental): Normal Saline IV with AD-cSVF cells
  Interventions: Procedure: Normal Saline IV

INTERVENTIONS:
Procedure: Lipoaspiration — Closed syringe harvesting subdermal fat
  Arms: Lipoaspiration Arm 1
Procedure: ADcSVF isolation — Isolation of AD-cSVF from lipoaspirate via enzymatic digestion
  Arms: AD-cSVF Arm 2
Procedure: Normal Saline IV — Normal Saline IV containing autologous AD-cSVF
  Arms: Normal Saline IV Arm 3

SUMMARY:
Reflex Sympathetic Dystrophy (RSD), Complex Regional Pain Syndrome (CRPS), Causalgia, and Fibromyalgia represent progressive systemic pain conditions which often worsen over time. They appear to be dysregulation of the central nervous system (CNS) and the autonomic system (sympathetic/parasympathetic) which cause extensive functional losses, impairment, and disabilities. They are often associated with injury sites (including surgical) which produce constant, often disabling pain and motor-sensory losses.

Treatments are often ineffective and include medications (often high dose opiates), Physical Therapy (PT), and surgical interventions (sympathectomy, ablation) or insertion stimulators of the CNS.

Study is an interventional study to document the safety and efficacy of use of adipose-derived cellular stromal vascular fraction (AD-cSVF) in chronic pain and dysfunction disease groups.

DETAILED DESCRIPTION:
Reflex Sympathetic Dystrophy (RSD), Complex Regional Pain Syndrome (CRPS), Causalgia, and Fibromyalgia represent progressive systemic pain conditions which often worsen over time. They appear to be dysregulation of the central nervous system (CNS) and the autonomic system (sympathetic/parasympathetic) which cause extensive functional losses, impairment, and disabilities. They are often associated with injury sites (including surgical) which produce constant, often disabling pain and motor-sensory losses.

Treatments are often ineffective and include medications (often high dose opiates), physical therapy (PT(, and surgical interventions (sympathectomy, ablation) or insertion stimulators of the CNS.

Clinical Features include neurogenic inflammation, nociceptive sensitization, vasomotor dysfunction and maladaptive neuroplasticity. As these often seem related to specific injury sites (trauma, surgical, etc.) which are followed with severe pain sensations such as stabbing, burning, throbbing, and local muscular spasms or hemiparesis. In addition, there are many reports of visual change, dropping attacks (sudden falling), joint soreness, and other systemic symptoms associated with potentially any organ in the body.

Diagnosis typically recognizes 3 distinct "types" which do not appear to be sequential in nature. Type 1 characterization is severe, burning sensory change near an injury site, musculoskeletal and joint stiffness. Type 2 demonstrates very high pain levels, swelling, muscular atrophy, joint degeneration, depression, and other concomitant dysfunctions. Type 3 features irreversible changes to skin/bone, and extreme loss of function of muscle (atrophic primarily) and tendons. A significant percentage (13-70 ) are felt to be at risk if neurological injuries, hemiplegia, enhanced vasomotor issues due to enhanced sympathetic actions and neurotransmission issues.

This study includes microcannula harvesting of subdermal adipose tissues, incubation, digestion and isolation of AD-cSVF. This stromal cellular pellet (without actual extracellular matrix or stromal elements) is then suspended in 500 cc sterile Normal Saline (NS) and deployed via peripheral intravenous route. Evaluations of safety issues are measured at intervals (both severe and non-severe categories) and by repeated pulmonary function studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of RSD, CRPS, and severe Fibromyalgia
* Ability to provide Informed Consent (or as parent or legal guardian)

Exclusion Criteria:

* Patients with severe comorbidities which, in opinion of PI or provider associates. would be unsafe or not advised to be able to comply with study or follow up requirements
* Patients with documented Opiate abuse
* Patient taking corticosteroid therapy, immune suppression, or chemotherapeutic regimen within 6 months of entry

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Adverse and Severe Adverse Reaction Report | 12 months
  Evaluate any Adverse or Severe Adverse Reactions

SECONDARY OUTCOMES:
Change from Baseline Pain Levels | 1 month, 6 month, 1 year
  Pain Scale Questionnaire 1-10
Change in Quality of Life from Baseline | 6 months, 12 months
  Quality of Life Questionnaire (QoL)
Change from Baseline of Lifestyle | 6 months, 12 months
  Fibromyalgia Impact Questionnaire (FIQR)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn C Terry, MD, Principal Investigator — Global Alliance for Regenerative Medicine (GARM)
Locations (2):
- Regenevita LLC, Stevensville, Montana, United States
- GARM, Roatán, Hn, Honduras

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartzman RJ, Erwin KL, Alexander GM. The natural history of complex regional pain syndrome. Clin J Pain. 2009 May;25(4):273-80. doi: 10.1097/AJP.0b013e31818ecea5. PMID 19590474
- [Background] Marinus J, Moseley GL, Birklein F, Baron R, Maihofner C, Kingery WS, van Hilten JJ. Clinical features and pathophysiology of complex regional pain syndrome. Lancet Neurol. 2011 Jul;10(7):637-48. doi: 10.1016/S1474-4422(11)70106-5. PMID 21683929
- [Background] Veldman PH, Reynen HM, Arntz IE, Goris RJ. Signs and symptoms of reflex sympathetic dystrophy: prospective study of 829 patients. Lancet. 1993 Oct 23;342(8878):1012-6. doi: 10.1016/0140-6736(93)92877-v. PMID 8105263
- [Background] Maihofner C, Forster C, Birklein F, Neundorfer B, Handwerker HO. Brain processing during mechanical hyperalgesia in complex regional pain syndrome: a functional MRI study. Pain. 2005 Mar;114(1-2):93-103. doi: 10.1016/j.pain.2004.12.001. Epub 2005 Jan 26. PMID 15733635
- [Background] Watkins LR, Maier SF. Immune regulation of central nervous system functions: from sickness responses to pathological pain. J Intern Med. 2005 Feb;257(2):139-55. doi: 10.1111/j.1365-2796.2004.01443.x. PMID 15656873
- [Background] Birklein F. Complex regional pain syndrome. J Neurol. 2005 Feb;252(2):131-8. doi: 10.1007/s00415-005-0737-8. PMID 15729516
- [Background] Lee BH, Scharff L, Sethna NF, McCarthy CF, Scott-Sutherland J, Shea AM, Sullivan P, Meier P, Zurakowski D, Masek BJ, Berde CB. Physical therapy and cognitive-behavioral treatment for complex regional pain syndromes. J Pediatr. 2002 Jul;141(1):135-40. doi: 10.1067/mpd.2002.124380. PMID 12091866
- [Background] van de Meent H, Oerlemans M, Bruggeman A, Klomp F, van Dongen R, Oostendorp R, Frolke JP. Safety of "pain exposure" physical therapy in patients with complex regional pain syndrome type 1. Pain. 2011 Jun;152(6):1431-1438. doi: 10.1016/j.pain.2011.02.032. Epub 2011 Apr 6. PMID 21474244
- [Background] Swart CM, Stins JF, Beek PJ. Cortical changes in complex regional pain syndrome (CRPS). Eur J Pain. 2009 Oct;13(9):902-7. doi: 10.1016/j.ejpain.2008.11.010. Epub 2008 Dec 19. PMID 19101181
- [Background] Chopra P, Cooper MS. Treatment of Complex Regional Pain Syndrome (CRPS) using low dose naltrexone (LDN). J Neuroimmune Pharmacol. 2013 Jun;8(3):470-6. doi: 10.1007/s11481-013-9451-y. Epub 2013 Apr 2. PMID 23546884
- [Background] Azari P, Lindsay DR, Briones D, Clarke C, Buchheit T, Pyati S. Efficacy and safety of ketamine in patients with complex regional pain syndrome: a systematic review. CNS Drugs. 2012 Mar 1;26(3):215-28. doi: 10.2165/11595200-000000000-00000. PMID 22136149
- [Background] Opal SM, Wiest PM, Olds GR. Traveler's diarrhea: methods of prevention and treatment. R I Med J (1976). 1990 May;73(5):199-204. PMID 2343234
- [Background] Varenna M, Adami S, Rossini M, Gatti D, Idolazzi L, Zucchi F, Malavolta N, Sinigaglia L. Treatment of complex regional pain syndrome type I with neridronate: a randomized, double-blind, placebo-controlled study. Rheumatology (Oxford). 2013 Mar;52(3):534-42. doi: 10.1093/rheumatology/kes312. Epub 2012 Nov 30. PMID 23204550
- [Background] Gainer MJ. Hypnotherapy for reflex sympathetic dystrophy. Am J Clin Hypn. 1992 Apr;34(4):227-32. doi: 10.1080/00029157.1992.10402852. PMID 1349789
- [Background] Hamdi TN. The Copeland intraocular lens: five to ten years later. Ophthalmology. 1979 Jun;86(6):984-96. doi: 10.1016/s0161-6420(79)35409-4. PMID 534104